CLINICAL TRIAL: NCT03377634
Title: A Mobile Intervention to Reduce Pain and Improve Health (MORPH) in Obese Older Adults
Brief Title: A Mobile Intervention to Reduce Pain and Improve Health (MORPH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00046364; 1R21AG058249-01 (NIH)
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain; Obesity; Sedentary Lifestyle
Keywords: Older Adults; Physical Activity; MORPH; Telecoaching; mHealth; Weight Loss; Sedentary Behavior; Pain; Design; RCT; Randomized Controlled Trial
MeSH Terms: conditions — Chronic Pain; Obesity; Sedentary Behavior; Motor Activity; Weight Loss; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants receive the MORPH intervention.
  Interventions: Behavioral: MORPH
- Control (No Intervention): The wait list control participants receive usual care and are offered intervention materials on completion of the study.

INTERVENTIONS:
Behavioral: MORPH — Participants will engage in 12 weekly group coaching sessions discussion behavioral approaches to pain management, weight loss, and daily physical activity. The first three sessions (i.e., weeks 1 - 3) will occur in-person, and the remaining 9 will take place via telephone. All intervention participants will receive access to an activity monitor, smart scale, and smartphone app that aims to provide support for daily physical activity and weight loss.
  Arms: Intervention

SUMMARY:
Chronic pain contributes to declining health and function in older adults; effects that are intensified by obesity and sedentary (sitting) behavior. The purpose of this study is to develop and test a novel, patient-centered intervention to reduce pain and improve physical function in older, obese adults. The study will utilize a combination of telephone based coaching and smartphone tools to deliver this novel intervention to decrease both body weight and sitting behavior. The long-term goals of this project are to test the efficacy of the intervention and to develop it as a tool for clinicians to provide outside-of-clinic patient-centered support for overweight/obese older adults with chronic pain.

DETAILED DESCRIPTION:
Chronic pain has emerged as an urgent age-related health issue that significantly effects physical functioning and quality of life, with the unfavorable effects worsened by both obesity and sedentary behavior. The annual cost of pain in the United States is nearly 30% higher than the combined costs of cancer and diabetes. In 2016, the NIH called for a National Pain Strategy to: 1) expand non-pharmacological treatment options in older adults, who are particularly susceptible to the side effects of opioid and other pain medications; 2) develop accessible treatments that are tailored to individuals; and 3) increase the development of self-management programs for chronic pain. The purpose of this R-21 is to develop and test the feasibility and acceptability of a novel, patient-centered intervention to reduce chronic pain and improve physical functioning in older adults, leveraging the combination of telecoaching and individually-adaptive mHealth tools to decrease both body mass and sedentary behavior. A pilot randomized controlled trial will be conducted to provide initial evidence for effect sizes (pain and physical function) associated with the proposed intervention, and to estimate the sample size needed for a full scale randomized controlled trial design that compares the effects of the intervention versus usual care on pain ratings and physical function in overweight/obese older adults with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Own smartphone
* Pain in 2 of 5 areas (i.e., back, neck, shoulders, hips, knees) on most days during the previous 3 months
* No contraindication for participation in exercise with approval for participation by their physician
* Obese (BMI=30-45 kg/m2)
* Weight-stable (i.e., no weight loss or gain > 5% in the past 6 months)
* Low-active (i.e., engaging in less than 2 days/week of structured physical activity for at least 20 minutes).
* Approved for participation by LMC Pain Center Director and Dr. Brooks
* Willingness to provide consent; Agree to all study procedures and assessments; Able to provide own transportation to study visits
* Access to home Wi-Fi and smartphone device

Exclusion Criteria:

* Dependent on cane or walker
* >1 fall (injurious or non-injurious) in past year
* Vision insufficient to read a smartphone screen, unable to read
* Participation in regular resistance training and/or > 20 mins/d of aerobic exercise in past 6 months
* No contraindication to exercise
* Unable to walk without assistive devices
* Cognitive impairment as indicated by a Montreal Cognitive Assessment score < 22
* Uncontrolled hypertension (>160/90 mmHg);
* Current or recent past (within 1 year) severe symptomatic heart disease, uncontrolled angina, stroke, chronic respiratory disease requiring oxygen, neurological or hematological disease; cancer requiring treatment in past yr, except non-melanoma skin cancers
* Regular use of: growth hormones, oral steroids, or prescription osteoporosis medications
* Current participation in other research study targeting pain, physical activity, or weight loss

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber K Brooks, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center Pain Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fanning J, Brooks AK, Ip E, Nicklas BJ, Rejeski WJ, Nesbit B, Ford S. A Mobile Health Behavior Intervention to Reduce Pain and Improve Health in Older Adults With Obesity and Chronic Pain: The MORPH Pilot Trial. Front Digit Health. 2020 Dec;2:598456. doi: 10.3389/fdgth.2020.598456. Epub 2020 Dec 18. PMID 33817686
- [Derived] Fanning J, Brooks AK, Ip E, Nicklas BJ, Rejeski WJ. A Mobile Health Intervention to Reduce Pain and Improve Health (MORPH) in Older Adults With Obesity: Protocol for the MORPH Trial. JMIR Res Protoc. 2018 May 14;7(5):e128. doi: 10.2196/resprot.9712. PMID 29759957

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five participants were assigned to an usability testing period. For the duration of this period, intervention staff kept detailed notation of software and usability challenges, and iterations were made according to information gathered from this period. Notably, these iterations do not affect the overarching structure of the intervention, but will ensure all components of the program are maximally usability for the older adult with chronic pain.
Period: Intervention Usability Testing Period
Arm/Group | Intervention | Control
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0
Period: Study Period
Arm/Group | Intervention | Control
Started (Data from this period does not include the 5 subjects from the usability period because outcome measure information was not collected from those five subjects.) | 15 | 13
Completed | 13 | 13
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.12 (5.43) | 70.32 (5.20) | 70.21 (5.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 12 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in PROMIS Pain Intensity Scale
Description: The Pain Intensity Scale tasks participants with rating how much they hurt on a scale of 1 (had no pain) to 5 (very severe). Final scores are given as T-scores, with higher scores representing worse intensity. PROMIS scores are a t-score representing relationships with an estimated population average collected on a general US sample of adults as well as clinical samples. On this t distribution, 50 represents the population average with a standard deviation of 10. Thus, a score of 55 represents a score that is a half-standard deviation about the US national average, and a 40 represents a score that is 1 standard deviation below the national average. Scores were computed using the HealthMeasures.org scoring service as recommended for PROMIS measures.
Time Frame: Baseline to 12 weeks
Population: Three subjects did not do follow up visits in the intervention arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 13
units on a scale | -8.08 (9.00) | -1.92 (5.71)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — Analysis of covariance on change in PROMIS Pain intensity, with group as fixed effect and controlling for baseline pain intensity; p = 0.11, ANCOVA

2. Primary Outcome: Change in PROMIS Pain Interference Scale
Description: The Pain Interference Scale captures the impact of pain on valued areas of an individual's life (e.g., how much did pain interfere with your day to day activities) on a scale of 1 (not at all) to 5 (very much). Final scores are given as T-scores, with higher scores representing worse interference. PROMIS scores are a t-score representing relationships with an estimated population average collected on a general US sample of adults as well as clinical samples. On this t distribution, 50 represents the population average with a standard deviation of 10. Thus, a score of 55 represents a score that is a half-standard deviation about the US national average, and a 40 represents a score that is 1 standard deviation below the national average. Scores were computed using the HealthMeasures.org scoring service as recommended for PROMIS measures.
Time Frame: Baseline to 12 weeks
Population: Three subjects did not do follow up visits in the intervention arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 13
units on a scale | 2.76 (10.54) | 3.11 (5.97)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — Analysis of covariance on change in PROMIS pain interference, with group as fixed effect and controlling for baseline pain interference; p = .99, ANCOVA

3. Primary Outcome: Change in Short Physical Performance Battery
Description: This test of lower-extremity function consists of 4-m walk at usual pace, a timed repeated chair stand, and 3 increasingly difficult standing balance tests. Each measure is assigned a categorical score ranging from 0 (inability to complete the test) to 4 (best performance) resulting in a final score of 0-12. Higher scores denotes better outcomes.
Time Frame: Baseline to 12 weeks
Population: Three subjects did not do follow up visits in the intervention arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 13
score on a scale | 0.67 (1.50) | 0.00 (1.0)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — Analysis of covariance on change in SPPB, with group as fixed effect and controlling for baseline SPPB; p = .14, ANCOVA

4. Secondary Outcome: Change in Weight
Description: Weight will be assessed weekly.
Time Frame: Baseline to 12 weeks
Population: One subject did not do follow up visits in the intervention arm.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 14 | 13
kg | -2.27 (4.34) | -0.18 (1.55)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — Analysis of covariance on change in weight, with group as fixed effect and controlling for baseline weight; p = .11, ANCOVA

5. Secondary Outcome: Activity Minutes
Description: Activity Minutes will be assessed using ActivPal activity monitors (PAL Technologies Ltd, Glasgow, UK) worn at the thigh for 7 consecutive days. We will assess (a) number of daily minutes spent in light-intensity physical activity as reported by the ActivPal (range: 0-1440, more minutes of light activity are favorable); (b) number of daily minutes spent in moderate-intensity physical activity as reported by the ActivPal (range: 0-1440, more minutes of moderate activity are favorable).
Time Frame: Baseline and Week 12
Population: Only 9 in each arm with 2+ days of valid data at each time point
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 9 | 9
minutes per day
  Baseline | 53 (23.57) | 73.35 (46.42)
  Week 12 | 51 (27.08) | 62.70 (35.53)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — Analysis of covariance on change in activity time, with group as fixed effect and controlling for baseline stepping time; p = .65, ANCOVA

6. Secondary Outcome: Sitting Time
Description: daily minutes of sedentary time as recorded on the ActivPALTM 4 device
Time Frame: Week 12
Population: Only 9 subjects had 2+ days of valid data at each time point
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 9 | 9
minutes per day
  baseline | 698.48 (123.29) | 642.12 (176.48)
  Week 12 | 682.26 (182.49) | 684.86 (154.92)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — Analysis of covariance on change in sitting time, with group as fixed effect and controlling for baseline sitting time; p = .41, ANCOVA

7. Secondary Outcome: Sit to Stand Transitions
Description: Transitions will be assessed using ActivPal activity monitors (PAL Technologies Ltd, Glasgow, UK) worn at the thigh for 7 consecutive days. We will assess number of daily transitions from sitting to non-sitting behavior, captured via the ActivPal inclinometer (range: 0 - infinity; a higher number of transitions are favorable).
Time Frame: Baseline and Week 13
Population: Only 9 subjects in each arm with 2+ days of valid data at each time point
Measure: Mean (Standard Deviation); unit: number of transitions per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 9 | 9
number of transitions per day
  baseline | 31.33 (10.20) | 36.44 (9.72)
  Week 12 | 29.22 (11.33) | 37.44 (10.55)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other — Analysis of covariance on change in sit to stand transitions, with group as fixed effect and controlling for baseline transitions; p = .28, ANCOVA

8. Secondary Outcome: Participant Retention
Description: The extent to which participants were retained in the study (minimum retention goal of 80%). The number of participants that complete the study over the number that were enrolled.
Time Frame: Baseline to 12 weeks
Population: Three lost to follow-up from intervention arm.
Measure: Number; unit: percentage of subjects completing
Arm/Group | Intervention | Control
Number analyzed (Participants) | 15 | 13
percentage of subjects completing | 80 | 100

9. Secondary Outcome: Utilization of Study Application
Description: The extent to which participants utilize the study application, as defined by an average weekly use of 7 application accesses per week for the duration of the study period.
Time Frame: Baseline to 12 weeks
Population: This outcome only pertains to the intervention arm.
Measure: Mean (Standard Deviation); unit: number of times accessing per week
Arm/Group | Intervention | Control
Number analyzed (Participants) | 15 | 0
number of times accessing per week | 10.84 (9.64) |

ADVERSE EVENTS:
Time Frame: Baseline through Week 12
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/13
Other Adverse Events (participants affected / at risk) | 6/15 | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=15) | Control (N=13)
small intestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=15) | Control (N=13)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Strep Throat (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT03377634/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT03377634/Prot_SAP_001.pdf